CLINICAL TRIAL: NCT05724290
Title: The Regulatory Mechanism of EGR2 Mediated by miR-150-5p on Allergic Rhinitis
Brief Title: Mechanism of EGR2 in Allergic Rhinitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zu-xia Ma (Other)
Responsible Party: Sponsor-Investigator, Zu-xia Ma, Professor, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: [2018]1182
Record Dates: First submitted 2023-02-07; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Rhinitis, Allergic
Keywords: nasal polyps; chronic rhinosinusitis; atopic NPs; non-atopic NPs; EGR2
MeSH Terms: conditions — Rhinitis, Allergic; Nasal Polyps

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immunohistochemistry (Experimental): Thirty-eight patients with confirmed nasal polyps (20 with primary CRSwNP and allergic rhinitis (AR) and 18 with CRSWNP) and 20 patients with chronic hypertrophic rhinitis were included. The nasal polyps and mucosal specimens of all patients were collected and analyzed by immunohistochemistry
  Interventions: Genetic: EGR2
- WestBlot (Experimental): Thirty-eight patients with confirmed nasal polyps (20 with primary CRSwNP and allergic rhinitis (AR) and 18 with CRSWNP) and 20 patients with chronic hypertrophic rhinitis were included. The nasal polyps and mucosal specimens of all patients were collected and analyzed by Western Blot.
  Interventions: Genetic: EGR2

INTERVENTIONS:
Genetic: EGR2 — We investigated the expression of EGR2 in patients with nasal polyps through immunohistochemistry.

SUMMARY:
EGR2 may be a target for the treatment of nasal polyps.

DETAILED DESCRIPTION:
There is much debate about the etiology of nasal polyps, so the pathogenesis of nasal polyps still needs to be clarified. Surgery for noninflammatory nasal polyps may be better control, but surgery is not effective for recurrent sinusitis and nasal polyps. Therefore, more research is needed to determine the best targeted therapy for nasal polyps. We found that EGR2 expression was upregulated in CRSwNP patients with allergic rhinitis.In addition, the expression of EGR2 in CRSwNP mucosa was significantly higher than that in the control group, and the expression of EGR2 in CRSwNP with allergic rhinitis was higher than that in CRSwNP without allergic rhinitis. EGR2 may be involved in the pathogenesis of nasal polyps, and may also be related to the severity and recurrence of nasal polyps. EGR2 may be a target for the treatment of nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

All patients were stopped by systemic or topical corticosteroid treatment at least one month before the study.

Exclusion Criteria:

Patients had NPs accompanied by choanal polyps, fungal nasal sinusitis, cystic fibrosis, acute upper airway upper infection or other systemic diseases.

Ages: 16 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-05-05 (Estimated)

PRIMARY OUTCOMES:
expression of EGR2 | one months
  expression of EGR2 were analyzed by immunohistochemistry and Western Blot

CONTACTS AND LOCATIONS:
Overall Officials: Yong Luo, Doctor, Principal Investigator — Zunyi Medical College
Locations (1):
- Department of Central Laboratory of the Third Affiliated Hospital of ZunYi Medical University, Zunyi, China

IPD SHARING:
Plan to Share IPD: No